CLINICAL TRIAL: NCT05680259
Title: Assessment of the Effects of Maela Connected Follow-up on Well-being and Pain After Lumbar Spine Surgery
Acronym: HOSPITEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0016
Record Dates: First submitted 2022-10-06; First posted 2023-01-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Spine Surgery; Quality of Life; Pain
Keywords: mobile app follow-up; lumbar spine surgery; Quality of Life; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maela connected follow-up (Experimental): patient will benefit of the Maela connected follow-up
  Interventions: Other: Maela connected follow-up
- control group (Active Comparator): control group with a traditional follow-up
  Interventions: Other: traditional follow-up

INTERVENTIONS:
Other: Maela connected follow-up — Measures of pain, quality of life and health related variables (coping, self-efficacy, beliefs about pain) will be done at four times before and after surgery.
  Arms: Maela connected follow-up
Other: traditional follow-up — medical recommendations and prescriptions at hospital discharge. Measures of pain, quality of life and health related variables (coping, self-efficacy, beliefs about pain) will be done at four times before and after surgery.
  Arms: control group

SUMMARY:
Digital technologies could reduce the length of hospital stay and improve post-operative recuperation after discharge by offering a remote follow-up. No study has investigated the effects of connected follow-up on lumbar spine inpatients.

The purpose of this project is to assess the effects of connected follow-up on pain and quality of life after lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* First ever lumbar spine surgery in the context of a degenerative spinal pathology
* Age between 18 and 60 yo
* Providing free and informed consent to participate
* Having a smartphone able to process MAELA application

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Variation of number of well-being patients in both groups | two months
  Variation of number of well-being patients in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No